CLINICAL TRIAL: NCT00802464
Title: Immunogenicity and Safety Study of Different Formulations of GSK Biologicals' Herpes Zoster Vaccine 1437173A When Administered Twice in Adults Aged 50 Years and Older
Brief Title: Immunogenicity and Safety Study of GSK Biologicals' Herpes Zoster Vaccine With Various Formulations in Adults >= 50 Years
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 112077; 2008-005120-86 (EudraCT Number)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2017-12-12 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Herpes Zoster
Keywords: Cytokine; Vaccine; Herpes Zoster (HZ); Cell mediated immunity (CMI); Antibody response; Varicella Zoster Virus (VZV); Shingles
MeSH Terms: conditions — Herpes Zoster; Chickenpox | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- GSK1437173A formulation 1 Group (Experimental): Male or female subjects, 50 years of age or above, who received 2 doses of GSK1437173A (gE/ASO1B and gE/ASO1E) formulation 1 vaccine, administered intramuscularly in the upper deltoid region of the non-dominant arm on a 0, 2 month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A
- GSK1437173A formulation 2 Group (Experimental): Male or female subjects, 50 years of age or above, who received 2 doses of GSK1437173A (gE/ASO1B and gE/ASO1E) GSK1437173A formulation 2 vaccine, administered intramuscularly in the upper deltoid region of the non-dominant arm on a 0, 2 month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A
- GSK1437173A formulation 3 Group (Experimental): Male or female subjects, 50 years of age or above, who received 2 doses of GSK1437173A (gE/ASO1B and gE/ASO1E) formulation 3 vaccine, administered intramuscularly in the upper deltoid region of the non-dominant arm on a 0, 2 month schedule.
  Interventions: Biological: Herpes zoster vaccine GSK1437173A
- Control Group (Placebo Comparator): Male or female subjects, 50 years of age or above, who received 2 doses of saline solution (placebo), administered intramuscularly in the upper deltoid region of the non-dominant arm on a 0, 2 month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Herpes zoster vaccine GSK1437173A — 2 vaccinations at Months 0 and 2 with GSK1437173A (different formulations)
  Other Names: gE/AS01E; gE/AS01B
  Arms: GSK1437173A formulation 1 Group; GSK1437173A formulation 2 Group; GSK1437173A formulation 3 Group
Biological: Placebo — 2 vaccinations at Months 0 and 2 with placebo
  Other Names: Placebo/Saline
  Arms: Control Group

SUMMARY:
The goal of this randomized observer-blind trial is to further refine the formulation of vaccines containing GSK1437173A in older adults by comparing the cellular and humoral immune responses and the safety profiles of the different formulations.

ELIGIBILITY:
Inclusion Criteria:

* A male or female 50 years of age or above at the time of the first vaccination;
* Written informed consent obtained from the subject;
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study;
* If the subject is female, she must be of non-childbearing potential, or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period;
* Chronic administration (defined as more than 14 consecutive days) of immunosuppressants or other immune-modifying drugs within three months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month before the first study vaccination or scheduled within 30 days after study vaccination;
* Previous vaccination against HZ;
* Previous vaccination against varicella;
* History of HZ;
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine;
* Any confirmed or suspected immunosuppressive or immunodeficient condition resulting from disease or immunosuppressive/cytotoxic therapy;
* Administration of immunoglobulins and/or any blood products within the 3 months preceding the first injection of study vaccine or planned administration during the study period;
* Acute disease at the time of enrolment.
* Any other condition that, in the opinion of the investigator, might interfere with the evaluations required by the study;
* History of or current drug and/or alcohol abuse;
* Pregnant or lactating female;
* Female planning to become pregnant or planning to discontinue contraceptive precautions if of childbearing potential.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2009-01-12 (Actual); Primary Completion 2010-07-02 (Actual); Study Completion 2010-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (11):
- United States (7):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Edison, New Jersey
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Pittsburgh, Pennsylvania
- GSK Investigational Site, Hradec Králové, Czechia
- Spain (3):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Mahadahonda( Madrid
  - GSK Investigational Site, Marid

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Chlibek R, Bayas JM, Collins H, de la Pinta ML, Ledent E, Mols JF, Heineman TC. Safety and immunogenicity of an AS01-adjuvanted varicella-zoster virus subunit candidate vaccine against herpes zoster in adults >=50 years of age. J Infect Dis. 2013 Dec 15;208(12):1953-61. doi: 10.1093/infdis/jit365. Epub 2013 Jul 31. PMID 23904292
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 112077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 112077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 112077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 112077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 112077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 112077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 112077 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Group: Male or female subjects, 50 years of age or above, who received 2 doses of saline solution (placebo), administered intramuscularly in the upper deltoid region of the non-dominant arm, on a 0, 2 month schedule.
- GSK1437173A Formulation 3 Group: Male or female subjects, 50 years of age or above, who received 2 doses of GSK1437173A (gE/AS01B and gE/AS01E) formulation 3 vaccine, administered intramuscularly in the upper deltoid region of the non-dominant arm, on a 0, 2 month schedule.
- GSK1437173A Formulation 2 Group: Male or female subjects, 50 years of age or above, who received 2 doses of GSK1437173A (gE/AS01B and gE/AS01E) formulation 2 vaccine, administered intramuscularly in the upper deltoid region of the non-dominant arm, on a 0, 2 month schedule.
- GSK1437173A Formulation 1 Group: Male or female subjects, 50 years of age or above, who received 2 doses of GSK1437173A (gE/AS01B and gE/AS01E) formulation 1 vaccine, administered intramuscularly in the upper deltoid region of the non-dominant arm, on a 0, 2 month schedule.
Period: Month 0 - Month 8
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Started | 38 | 73 | 149 | 150
Completed | 38 | 70 | 142 | 141
Not Completed | 0 | 3 | 7 | 9
Not completed — Adverse Event | 0 | 1 | 1 | 2
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 5
Not completed — Lost to Follow-up | 0 | 1 | 2 | 2
Not completed — Other | 0 | 0 | 1 | 0
Period: Month 8 - Month 14
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Started | 34 | 65 | 130 | 126
Completed | 33 | 63 | 129 | 126
Not Completed | 1 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group | Total
Number analyzed (Participants) | 38 | 73 | 149 | 150 | 410
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.0 (9.0) | 65.1 (8.7) | 65.1 (9.9) | 65.0 (8.9) | 65.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 40 | 89 | 81 | 232
  Male | 16 | 33 | 60 | 69 | 178
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African Heritage / African American | 0 | 1 | 2 | 6 | 9
  Race/Ethnicity: American Indian or Alaskan Native | 0 | 0 | 1 | 2 | 3
  Race/Ethnicity: Other | 0 | 0 | 0 | 1 | 1
  Race/Ethnicity: White - Arabic / North African Heritage | 0 | 0 | 1 | 0 | 1
  Race/Ethnicity: White - Caucasian / European Heritage | 38 | 72 | 145 | 141 | 396

OUTCOME MEASURES:

1. Primary Outcome: Frequency of gE-specific Cluster of Differentiation 4 (CD4+) T-cells Expressing at Least 2 Different Immunological Activation Markers
Description: The analysis focused on CD4+ T-cells expressing at least 2 immunological activation markers among Interferon gamma (IFN-γ), Interleukin 2 (IL-2), Tumour Necrosis Factor alpha (TNF-α) and CD40 Ligand (CD40L). Frequencies were determined by in vitro Intracellular Cytokine Staining (ICS).
Time Frame: One month after the second vaccination (Month 3)
Population: The analyses were performed on the According-to-Protocol (ATP) Cohort for immunogenicity, which included all evaluable subjects from Month 0 to 3. This included those subjects who met all eligibility criteria, complied with the protocol, with no elimination criteria during this part of the study and for whom immunogenicity measures were available.
Measure: Mean (Standard Deviation); unit: gE-specific CD4+ T-cells/million T-cells
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 32 | 70 | 126 | 125
gE-specific CD4+ T-cells/million T-cells | 231.82 (411.84) | 570.36 (610.10) | 2172.37 (1805.51) | 2582.80 (2154.92)
Statistical Analysis 1: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 1 Group; Fold increase in frequency of gE-specific CD4+ T-cells secreting at least 2 different immunological activation markers among IFN-γ, IL-2, TNF-α and CD40L for GSK1437173A Formulation 1 over GSK1437173A Formulation 3 Group; Test type: Other; Fold increase = 5.21, 95% CI 2-sided [3.89 to 6.98]
Statistical Analysis 2: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 2 Group; Fold increase in frequency of gE-specific CD4+ T-cells secreting at least 2 different immunological activation markers among IFN-γ, IL-2, TNF-α and CD40L for GSK1437173A Formulation 2 over GSK1437173A Formulation 3 Group; Test type: Other; Fold increase = 4.02, 95% CI 2-sided [3 to 5.4]
Statistical Analysis 3: Comparison: GSK1437173A Formulation 2 Group vs GSK1437173A Formulation 1 Group; Fold increase in frequency of gE-specific CD4+ T-cells secreting at least 2 different immunological activation markers among IFN-γ, IL-2, TNF-α and CD40L for GSK1437173A Formulation 1 over GSK1437173A Formulation 2 Group; Test type: Other; Fold increase = 1.3, 95% CI 2-sided [1.07 to 1.58]

2. Primary Outcome: Frequency of Varicella-Zoster Virus (VZV)-Specific CD4+ T-cells Expressing at Least 2 Different Immunological Activation Markers
Description: as for outcome 1
Time Frame: One month after the second vaccination (Month 3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: VZV-specific CD4+ T-cells/million T-cell
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 32 | 70 | 126 | 125
VZV-specific CD4+ T-cells/million T-cell | 457.43 (275.25) | 523.12 (396.01) | 1093.08 (927.18) | 1270.79 (1106.45)
Statistical Analysis 1: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 1 Group; [analysis description as in outcome 1, analysis 1]; Test type: Other; Fold increase = 2.12, 95% CI 2-sided [1.67 to 2.69]
Statistical Analysis 2: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 2 Group; [analysis description as in outcome 1, analysis 2]; Test type: Other; Fold increase = 1.63, 95% CI 2-sided [1.28 to 2.07]
Statistical Analysis 3: Comparison: GSK1437173A Formulation 2 Group vs GSK1437173A Formulation 1 Group; [analysis description as in outcome 1, analysis 3]; Test type: Other; Fold increase = 1.3, 95% CI 2-sided [1.09 to 1.56]

3. Primary Outcome: Anti-glycoprotein E (gE) Antibody Concentrations
Description: Concentrations were determined by enzyme-linked immunosorbent assay (ELISA) and are presented as geometric mean concentrations (GMCs), expressed in milli-international units per milliliter (mIU/mL).
Time Frame: One month after the second vaccination (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 36 | 70 | 133 | 132
mIU/mL | 1987.0 [1405.8 to 2808.6] | 14627.6 [11347.9 to 18855.1] | 49531.5 [44269.3 to 55419.2] | 68798.2 [61596.8 to 76841.5]
Statistical Analysis 1: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 1 Group; Fold increase in anti-gE antibody concentrations for GSK1437173A Formulation 1 Group over GSK1437173A Formulation 3 Group; Test type: Other; Fold increase = 4.72, 95% CI 2-sided [3.81 to 5.85]
Statistical Analysis 2: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 2 Group; Fold increase in anti-gE antibody concentrations for GSK1437173A Formulation 2 Group over GSK1437173A Formulation 3 Group; Test type: Other; Fold increase = 3.36, 95% CI 2-sided [2.72 to 4.17]
Statistical Analysis 3: Comparison: GSK1437173A Formulation 2 Group vs GSK1437173A Formulation 1 Group; Fold increase in anti-gE antibody concentrations for GSK1437173A Formulation 1 Group over GSK1437173A Formulation 2 Group; Test type: Other; Fold increase = 1.4, 95% CI 2-sided [1.17 to 1.68]

4. Primary Outcome: Anti-VZV Antibody Concentrations
Description: as for outcome 3
Time Frame: One month after the second vaccination (Month 3)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 36 | 70 | 133 | 132
mIU/mL | 1423.2 [1097.8 to 1845.0] | 2786.4 [2445.1 to 3175.3] | 4565.4 [4357.0 to 4783.7] | 4972.8 [4802.7 to 5148.8]
Statistical Analysis 1: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 1 Group; [analysis description as in outcome 3, analysis 1]; Test type: Other; Fold increase = 3.21, 36% CI 2-sided [2.64 to 3.9]
Statistical Analysis 2: Comparison: GSK1437173A Formulation 3 Group vs GSK1437173A Formulation 2 Group; [analysis description as in outcome 3, analysis 2]; Test type: Other; Fold increase = 2.44, 95% CI 2-sided [2.02 to 2.97]
Statistical Analysis 3: Comparison: GSK1437173A Formulation 2 Group vs GSK1437173A Formulation 1 Group; [analysis description as in outcome 3, analysis 3]; Test type: Other; Fold increase = 1.31, 95% CI 2-sided [1.12 to 1.54]

5. Secondary Outcome: Frequencies of gE-specific CD4+ T-cells Expressing at Least 2 Different Immunological Activation Markers
Description: as for outcome 1
Time Frame: At Month 0 and at Month 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gE-specific CD4+ T-cells/million T-cells
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 35 | 70 | 132 | 133
gE-specific CD4+ T-cells/million T-cells
  Month 0: number analyzed (Participants) | 35 | 65 | 132 | 133
  Month 0 | 210.18 (363.37) | 130.98 (115.90) | 196.52 (217.94) | 173.48 (203.54)
  Month 2: number analyzed (Participants) | 33 | 70 | 126 | 127
  Month 2 | 185.59 (310.06) | 189.46 (188.80) | 463.79 (386.94) | 430.50 (323.88)

6. Secondary Outcome: Frequency of VZV-specific CD4+ T-cells Expressing at Least 2 Different Immunological Activation Markers
Description: as for outcome 1
Time Frame: At Month 0 and at Month 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: VZV-specific CD4+ T-cells/million T-cell
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 35 | 68 | 131 | 133
VZV-specific CD4+ T-cells/million T-cell
  Month 0: number analyzed (Participants) | 35 | 65 | 131 | 133
  Month 0 | 533.97 (422.46) | 352.71 (283.42) | 457.28 (402.04) | 482.63 (512.05)
  Month 2: number analyzed (Participants) | 33 | 68 | 124 | 127
  Month 2 | 491.12 (330.34) | 410.69 (356.65) | 595.10 (588.51) | 574.54 (586.85)

7. Secondary Outcome: Anti-gE Antibody Concentrations
Description: as for outcome 3
Time Frame: At Month 0 and at Month 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 37 | 71 | 137 | 140
mIU/mL
  Month 0 | 1907.7 [1374.9 to 2646.9] | 1640.3 [1307.9 to 2057.3] | 1526.7 [1306.6 to 1783.8] | 1398.3 [1212.6 to 1612.5]
  Month 2: number analyzed (Participants) | 37 | 70 | 134 | 133
  Month 2 | 2022.3 [1484.6 to 2754.7] | 10022.8 [7593.7 to 13228.7] | 19962.3 [16894.4 to 23587.3] | 23942.4 [20536.9 to 27912.6]

8. Secondary Outcome: Anti-VZV Antibody Concentrations
Description: as for outcome 3
Time Frame: At Month 0 and at Month 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 37 | 71 | 137 | 140
mIU/mL
  Month 0 | 1505.5 [1191.7 to 1901.9] | 1289.6 [1100.3 to 1511.6] | 1215.9 [1077.4 to 1372.2] | 1175.8 [1051.0 to 1315.5]
  Month 2: number analyzed (Participants) | 37 | 70 | 134 | 133
  Month 2 | 1365.5 [1074.4 to 1735.4] | 2392.8 [2074.8 to 2759.5] | 3125.6 [2902.8 to 3365.5] | 3355.1 [3110.6 to 3618.9]

9. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-vaccination period after each dose and across doses
Population: The analyses were performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented, who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 38 | 73 | 149 | 150
Participants
  Any Pain, Dose 1 | 1 | 8 | 89 | 112
  Grade 3 Pain, Dose 1 | 0 | 0 | 1 | 0
  Any Redness, Dose 1 | 0 | 0 | 15 | 26
  Grade 3 Redness, Dose 1 | 0 | 0 | 2 | 2
  Any Swelling, Dose 1 | 0 | 1 | 9 | 8
  Grade 3 Swelling, Dose 1 | 0 | 0 | 1 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Pain, Dose 2 | 2 | 9 | 82 | 106
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Pain, Dose 2 | 0 | 0 | 1 | 6
  Any Redness, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Redness, Dose 2 | 0 | 3 | 19 | 37
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Redness, Dose 2 | 0 | 0 | 1 | 1
  Any Swelling, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Swelling, Dose 2 | 0 | 2 | 20 | 18
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 1
  Any Pain, Across Doses | 3 | 14 | 104 | 125
  Grade 3 Pain, Across Doses | 0 | 0 | 2 | 6
  Any Redness, Across Doses | 0 | 3 | 26 | 44
  Grade 3 Redness, Across Doses | 0 | 0 | 3 | 2
  Any Swelling, Across Doses | 0 | 3 | 25 | 23
  Grade 3 Swelling, Across Doses | 0 | 0 | 1 | 1

10. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms.
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms, headache, myalgia and fever [defined as axillary temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever higher than (>) 39.0 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: During the 7-day (Days 0-6)post-vaccination period after each dose and across doses
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 38 | 73 | 149 | 150
Participants
  Any Fatigue, Dose 1 | 3 | 10 | 32 | 42
  Grade 3 Fatigue, Dose 1 | 0 | 1 | 2 | 2
  Related Fatigue, Dose 1 | 3 | 9 | 28 | 39
  Any Gastr. sympt., Dose 1 | 1 | 1 | 10 | 8
  Grade 3 Gastr. sympt., Dose 1 | 1 | 0 | 2 | 0
  Related Gastr. sympt., Dose 1 | 0 | 0 | 7 | 7
  Any Headache, Dose 1 | 2 | 8 | 22 | 32
  Grade 3 Headache, Dose 1 | 0 | 0 | 0 | 1
  Related Headache, Dose 1 | 1 | 5 | 14 | 29
  Any Myalgia, Dose 1 | 1 | 8 | 36 | 42
  Grade 3 Myalgia, Dose 1 | 0 | 0 | 0 | 2
  Related Myalgia, Dose 1 | 1 | 6 | 29 | 40
  Any Temperature, Dose 1 | 0 | 0 | 7 | 11
  Grade 3 Temperature, Dose 1 | 0 | 0 | 0 | 0
  Related Temperature, Dose 1 | 0 | 0 | 3 | 8
  Any Fatigue, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Fatigue, Dose 2 | 5 | 10 | 41 | 58
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Fatigue, Dose 2 | 1 | 1 | 3 | 7
  Related Fatigue, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Related Fatigue, Dose 2 | 3 | 9 | 34 | 56
  Any Gastr. sympt., Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Gastr. sympt., Dose 2 | 2 | 4 | 12 | 12
  Grade 3 Gastr. sympt., Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Gastr. sympt., Dose 2 | 0 | 0 | 0 | 0
  Related Gastr. sympt., Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Related Gastr. sympt., Dose 2 | 1 | 3 | 8 | 9
  Any Headache, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Headache, Dose 2 | 3 | 5 | 25 | 42
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Headache, Dose 2 | 0 | 0 | 0 | 4
  Related Headache, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Related Headache, Dose 2 | 1 | 5 | 20 | 38
  Any Myalgia, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Myalgia, Dose 2 | 2 | 8 | 33 | 49
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Myalgia, Dose 2 | 1 | 0 | 2 | 6
  Related Myalgia, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Related Myalgia, Dose 2 | 2 | 8 | 26 | 48
  Any Temperature, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Any Temperature, Dose 2 | 1 | 0 | 14 | 21
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Grade 3 Temperature, Dose 2 | 0 | 0 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 37 | 72 | 143 | 143
  Related Temperature, Dose 2 | 1 | 0 | 11 | 20
  Any Fatigue, Across Doses | 7 | 16 | 52 | 72
  Grade 3 Fatigue, Across Doses | 1 | 2 | 5 | 9
  Related Fatigue, Across Doses | 6 | 14 | 45 | 71
  Any Gastr. sympt., Across Doses | 3 | 5 | 18 | 17
  Grade 3 Gastr. sympt., Across Doses | 1 | 0 | 2 | 0
  Related Gastr. sympt., Across Doses | 1 | 3 | 12 | 15
  Any Headache, Across Doses | 4 | 10 | 37 | 56
  Grade 3 Headache, Across Doses | 0 | 0 | 0 | 5
  Related Headache, Across Doses | 2 | 8 | 29 | 53
  Any Myalgia, Across Doses | 2 | 12 | 49 | 62
  Grade 3 Myalgia, Across Doses | 1 | 0 | 2 | 7
  Related Myalgia, Across Doses | 2 | 11 | 41 | 62
  Any Temperature, Across Doses | 1 | 0 | 18 | 25
  Grade 3 Temperature, Across Doses | 0 | 0 | 0 | 0
  Related Temperature, Across Doses | 1 | 0 | 13 | 23

11. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: Within the 30-day (Days 0-29) post-vaccination period
Population: The analyses were performed on the Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 38 | 73 | 149 | 150
Participants
  Any AE(s) | 6 | 18 | 37 | 46
  Grade 3 AE(s) | 1 | 1 | 3 | 5
  Related AE(s) | 0 | 2 | 15 | 24

12. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Month 0 up to Month 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 38 | 73 | 149 | 150
Participants
  Up to Month 3 | 2 | 3 | 4 | 4
  After Month 3 up to Month 8 | 1 | 4 | 2 | 2

13. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: as for outcome 12
Time Frame: During the period after Month 8 up to the end of the study at Month 14
Population: The analyses were performed on the Total Vaccinated Cohort for the Safety Follow-up (SFU) Month 14, which included all vaccinated subjects who were not withdrawn from the study during the period up to Month 3 nor from the SFU Month 8, and who signed the supplementary informed consent for participating to the End of study telephone contact.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 34 | 65 | 130 | 126
Participants | 1 | 3 | 1 | 4

14. Secondary Outcome: Number of Subjects With Any New Onset of Autoimmune Diseases (NOADs)
Description: Any new onset of autoimmune diseases were to be reported throughout the entire study period, whether or not they were considered to be possibly related to the treatment administration. These included neurological/demyelinating events, rheumatic and connective diseases, autoimmune endocrine diseases, inflammatory bowel diseases, autoimmune blood disorders, inflammatory skin disorders, other autoimmune/inflammatory events, autoimmune bullous skin diseases, vasculitis and liver autoimmune diseases.
Time Frame: From Month 0 until Month 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 38 | 73 | 149 | 150
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Number of Subjects With Any New Onset of Autoimmune Diseases (NOADs)
Description: as for outcome 14
Time Frame: During the period after Month 8 up to the end of the study at Month 14
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 34 | 65 | 130 | 126
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Subjects With Suspected Cases of Herpes Zoster (HZ)
Description: A suspected case of HZ was defined as a rash consistent with HZ.
Time Frame: From Month 0 until Month 8
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 38 | 73 | 149 | 150
Participants | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Subjects With Suspected Cases of Herpes Zoster (HZ)
Description: A suspected case of HZ is defined as a rash consistent with HZ.
Time Frame: During the period after Month 8 up to the end of the study at Month 14
Population: as for outcome 13
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
Number analyzed (Participants) | 34 | 65 | 130 | 126
Participants | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Subjects With Haematological and Biochemical Parameters Unknown, Below, Within or Above the Normal Ranges
Description: Hematological and biochemical parameters assessed were Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST), Basophils (BAS), Calcium (CAL), Creatinine (CREA), Eosinophils (EOS), Fibrinogen (FIBR), Hematocrit (HCT), Hemoglobin (HGB), Lactate Dehydrogenase (LDH), Lymphocytes (LYM), Mean Corpuscular Volume (MCV), Monocytes (MON), Neutrophils (NEU), Partial Thromboplastin Time (PTT), Platelets (PLAT), Prothrombin Time (PT), Red Blood Cells (RBC), Total Protein (TP) and White Blood Cells (WBC).
Time Frame: At Month 0
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 1 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 3 Group
Number analyzed (Participants) | 38 | 150 | 149 | 73
Participants
  ALT: Unknown | 0 | 0 | 0 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 35 | 146 | 142 | 71
  ALT: Above | 3 | 4 | 7 | 2
  AST: Unknown | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 38 | 148 | 146 | 71
  AST: Above | 0 | 2 | 3 | 2
  BAS: Unknown | 1 | 2 | 1 | 0
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 37 | 148 | 148 | 73
  BAS: Above | 0 | 0 | 0 | 0
  CAL: Unknown | 0 | 0 | 0 | 0
  CAL: Below | 0 | 0 | 0 | 0
  CAL: Normal | 38 | 150 | 144 | 73
  CAL: Above | 0 | 0 | 5 | 0
  CREA: Unknown | 0 | 0 | 0 | 0
  CREA: Below | 0 | 0 | 0 | 0
  CREA: Normal | 36 | 144 | 142 | 70
  CREA: Above | 2 | 6 | 7 | 3
  EOS: Unknown | 1 | 2 | 1 | 0
  EOS: Below | 0 | 11 | 12 | 8
  EOS: Normal | 36 | 132 | 135 | 65
  EOS: Above | 1 | 5 | 1 | 0
  FIBR: Unknown | 0 | 3 | 2 | 1
  FIBR: Below | 1 | 2 | 3 | 0
  FIBR: Normal | 34 | 127 | 126 | 56
  FIBR: Above | 3 | 18 | 18 | 16
  HCT: Unknown | 1 | 2 | 1 | 0
  HCT: Below | 2 | 12 | 9 | 1
  HCT: Normal | 35 | 135 | 135 | 71
  HCT: Above | 0 | 1 | 4 | 1
  HGB: Unknown | 1 | 2 | 1 | 0
  HGB: Below | 1 | 6 | 7 | 1
  HGB: Normal | 36 | 141 | 137 | 70
  HGB: Above | 0 | 1 | 4 | 2
  LDH: Unknown | 0 | 0 | 0 | 0
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 38 | 149 | 149 | 73
  LDH: Above | 0 | 1 | 0 | 0
  LYM: Unknown | 1 | 2 | 1 | 0
  LYM: Below | 1 | 2 | 1 | 1
  LYM: Normal | 35 | 146 | 145 | 72
  LYM: Above | 1 | 0 | 2 | 0
  MCV: Unknown | 1 | 2 | 1 | 0
  MCV: Below | 0 | 5 | 1 | 2
  MCV: Normal | 37 | 140 | 145 | 69
  MCV: Above | 0 | 3 | 2 | 2
  MON: Unknown | 1 | 2 | 1 | 0
  MON: Below | 1 | 6 | 4 | 2
  MON: Normal | 36 | 142 | 144 | 71
  MON: Above | 0 | 0 | 0 | 0
  NEU: Unknown | 1 | 2 | 1 | 0
  NEU: Below | 0 | 3 | 0 | 0
  NEU: Normal | 37 | 142 | 146 | 71
  NEU: Above | 0 | 3 | 2 | 2
  PTT: Unknown | 0 | 4 | 2 | 1
  PTT: Below | 1 | 10 | 5 | 1
  PTT: Normal | 36 | 135 | 137 | 70
  PTT: Above | 1 | 1 | 5 | 1
  PLAT: Unknown | 2 | 2 | 2 | 0
  PLAT: Below | 0 | 3 | 3 | 1
  PLAT: Normal | 35 | 144 | 143 | 70
  PLAT: Above | 1 | 1 | 1 | 2
  PT: Unknown | 0 | 4 | 2 | 1
  PT: Below | 2 | 7 | 2 | 3
  PT: Normal | 35 | 135 | 137 | 67
  PT: Above | 1 | 4 | 8 | 2
  RBC: Unknown | 1 | 2 | 1 | 0
  RBC: Below | 0 | 7 | 4 | 2
  RBC: Normal | 37 | 141 | 142 | 68
  RBC: Above | 0 | 0 | 2 | 3
  TP: Unknown | 0 | 0 | 0 | 0
  TP: Below | 0 | 0 | 0 | 0
  TP: Normal | 38 | 149 | 148 | 73
  TP: Above | 0 | 1 | 1 | 0
  WBC: Unknown | 1 | 2 | 1 | 0
  WBC: Below | 0 | 1 | 0 | 1
  WBC: Normal | 37 | 145 | 140 | 70
  WBC: Above | 0 | 2 | 8 | 2

19. Secondary Outcome: Number of Subjects With Haematological and Biochemical Parameters Unknown, Below, Within or Above the Normal Ranges
Description: as for outcome 18
Time Frame: At Month 2
Population: The analyses were performed on the Month 2 Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and who completed the Month 2 study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 1 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 3 Group
Number analyzed (Participants) | 38 | 143 | 144 | 72
Participants
  ALT: Unknown | 0 | 0 | 0 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 36 | 139 | 138 | 68
  ALT: Above | 2 | 4 | 6 | 4
  AST: Unknown | 0 | 0 | 0 | 1
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 38 | 139 | 140 | 67
  AST: Above | 0 | 4 | 4 | 4
  BAS: Unknown | 1 | 3 | 2 | 2
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 37 | 140 | 142 | 70
  BAS: Above | 0 | 0 | 0 | 0
  CAL: Unknown | 0 | 0 | 0 | 1
  CAL: Below | 0 | 2 | 1 | 0
  CAL: Normal | 38 | 137 | 136 | 71
  CAL: Above | 0 | 4 | 7 | 0
  CREA: Unknown | 0 | 0 | 0 | 1
  CREA: Below | 0 | 0 | 0 | 0
  CREA: Normal | 37 | 138 | 138 | 67
  CREA: Above | 1 | 5 | 6 | 4
  EOS: Unknown | 1 | 3 | 2 | 2
  EOS: Below | 1 | 12 | 12 | 7
  EOS: Normal | 35 | 125 | 129 | 62
  EOS: Above | 1 | 3 | 1 | 1
  FIBR: Unknown | 0 | 2 | 3 | 0
  FIBR: Below | 1 | 12 | 4 | 9
  FIBR: Normal | 34 | 124 | 131 | 59
  FIBR: Above | 3 | 5 | 6 | 4
  HCT: Unknown | 1 | 3 | 2 | 1
  HCT: Below | 2 | 12 | 11 | 4
  HCT: Normal | 35 | 126 | 126 | 65
  HCT: Above | 0 | 2 | 5 | 2
  HGB: Unknown | 1 | 3 | 2 | 1
  HGB: Below | 1 | 9 | 7 | 3
  HGB: Normal | 35 | 129 | 134 | 66
  HGB: Above | 1 | 2 | 1 | 2
  LDH: Unknown | 0 | 0 | 0 | 0
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 38 | 143 | 144 | 71
  LDH: Above | 0 | 0 | 0 | 1
  LYM: Unknown | 1 | 3 | 2 | 2
  LYM: Below | 0 | 2 | 2 | 3
  LYM: Normal | 37 | 137 | 139 | 67
  LYM: Above | 0 | 1 | 1 | 0
  MCV: Unknown | 1 | 3 | 2 | 1
  MCV: Below | 0 | 2 | 1 | 3
  MCV: Normal | 37 | 134 | 139 | 67
  MCV: Above | 0 | 4 | 2 | 1
  MON: Unknown | 1 | 3 | 2 | 2
  MON: Below | 3 | 10 | 9 | 6
  MON: Normal | 34 | 130 | 133 | 64
  MON: Above | 0 | 0 | 0 | 0
  NEU: Unknown | 1 | 3 | 2 | 2
  NEU: Below | 1 | 3 | 1 | 1
  NEU: Normal | 36 | 136 | 138 | 68
  NEU: Above | 0 | 1 | 3 | 1
  PTT: Unknown | 0 | 2 | 3 | 0
  PTT: Below | 0 | 1 | 1 | 0
  PTT: Normal | 37 | 132 | 129 | 64
  PTT: Above | 1 | 8 | 11 | 8
  PLAT: Unknown | 1 | 3 | 4 | 2
  PLAT: Below | 1 | 3 | 5 | 0
  PLAT: Normal | 36 | 137 | 135 | 68
  PLAT: Above | 0 | 0 | 0 | 2
  PT: Unknown | 0 | 2 | 3 | 0
  PT: Below | 0 | 0 | 1 | 0
  PT: Normal | 37 | 136 | 132 | 67
  PT: Above | 1 | 5 | 8 | 5
  RBC: Unknown | 1 | 3 | 2 | 1
  RBC: Below | 1 | 8 | 10 | 3
  RBC: Normal | 36 | 131 | 131 | 66
  RBC: Above | 0 | 1 | 1 | 2
  TP: Unknown | 0 | 0 | 0 | 0
  TP: Below | 0 | 1 | 0 | 0
  TP: Normal | 38 | 142 | 144 | 72
  TP: Above | 0 | 0 | 0 | 0
  WBC: Unknown | 1 | 3 | 2 | 2
  WBC: Below | 1 | 6 | 0 | 1
  WBC: Normal | 35 | 133 | 139 | 67
  WBC: Above | 1 | 1 | 3 | 2

20. Secondary Outcome: Number of Subjects With Haematological and Biochemical Parameters Unknown, Below, Within or Above the Normal Ranges
Description: as for outcome 18
Time Frame: At Month 3
Population: The analyses were performed on the Month 3 Total Vaccinated Cohort, which included all subjects with at least one vaccine administration documented and who completed the Month 3 study visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Group | GSK1437173A Formulation 1 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 3 Group
Number analyzed (Participants) | 38 | 142 | 142 | 72
Participants
  ALT: Unknown | 0 | 0 | 0 | 0
  ALT: Below | 0 | 0 | 0 | 0
  ALT: Normal | 36 | 138 | 139 | 70
  ALT: Above | 2 | 4 | 3 | 2
  AST: Unknown | 0 | 0 | 0 | 0
  AST: Below | 0 | 0 | 0 | 0
  AST: Normal | 38 | 139 | 140 | 70
  AST: Above | 0 | 3 | 2 | 2
  BAS: Unknown | 0 | 3 | 3 | 3
  BAS: Below | 0 | 0 | 0 | 0
  BAS: Normal | 38 | 139 | 139 | 69
  BAS: Above | 0 | 0 | 0 | 0
  CAL: Unknown | 0 | 0 | 0 | 0
  CAL: Below | 0 | 1 | 0 | 1
  CAL: Normal | 38 | 140 | 138 | 71
  CAL: Above | 0 | 1 | 4 | 0
  CREA: Unknown | 0 | 0 | 0 | 0
  CREA: Below | 0 | 0 | 0 | 0
  CREA: Normal | 37 | 135 | 134 | 68
  CREA: Above | 1 | 7 | 8 | 4
  EOS: Unknown | 0 | 3 | 3 | 3
  EOS: Below | 1 | 7 | 13 | 11
  EOS: Normal | 36 | 131 | 122 | 57
  EOS: Above | 1 | 1 | 4 | 1
  FIBR: Unknown | 0 | 3 | 0 | 2
  FIBR: Below | 1 | 5 | 4 | 2
  FIBR: Normal | 35 | 125 | 133 | 61
  FIBR: Above | 2 | 9 | 5 | 7
  HCT: Unknown | 0 | 3 | 3 | 4
  HCT: Below | 4 | 12 | 10 | 6
  HCT: Normal | 34 | 126 | 126 | 61
  HCT: Above | 0 | 1 | 3 | 1
  HGB: Unknown | 0 | 3 | 3 | 3
  HGB: Below | 2 | 10 | 5 | 3
  HGB: Normal | 35 | 127 | 133 | 65
  HGB: Above | 1 | 2 | 1 | 1
  LDH: Unknown | 0 | 0 | 0 | 0
  LDH: Below | 0 | 0 | 0 | 0
  LDH: Normal | 38 | 141 | 142 | 71
  LDH: Above | 0 | 1 | 0 | 1
  LYM: Unknown | 0 | 3 | 3 | 3
  LYM: Below | 0 | 3 | 2 | 1
  LYM: Normal | 38 | 136 | 136 | 68
  LYM: Above | 0 | 0 | 1 | 0
  MCV: Unknown | 0 | 3 | 3 | 4
  MCV: Below | 0 | 3 | 1 | 4
  MCV: Normal | 38 | 133 | 137 | 63
  MCV: Above | 0 | 3 | 1 | 1
  MON: Unknown | 0 | 3 | 3 | 3
  MON: Below | 0 | 9 | 13 | 8
  MON: Normal | 38 | 130 | 126 | 61
  MON: Above | 0 | 0 | 0 | 0
  NEU: Unknown | 0 | 3 | 3 | 3
  NEU: Below | 0 | 4 | 0 | 0
  NEU: Normal | 38 | 135 | 138 | 65
  NEU: Above | 0 | 0 | 1 | 4
  PTT: Unknown | 0 | 3 | 0 | 2
  PTT: Below | 0 | 0 | 0 | 0
  PTT: Normal | 37 | 131 | 136 | 68
  PTT: Above | 1 | 8 | 6 | 2
  PLAT: Unknown | 1 | 7 | 3 | 4
  PLAT: Below | 0 | 4 | 4 | 1
  PLAT: Normal | 37 | 131 | 134 | 66
  PLAT: Above | 0 | 0 | 1 | 1
  PT: Unknown | 0 | 3 | 0 | 2
  PT: Below | 0 | 0 | 0 | 0
  PT: Normal | 37 | 131 | 137 | 68
  PT: Above | 1 | 8 | 5 | 2
  RBC: Unknown | 0 | 3 | 3 | 4
  RBC: Below | 2 | 7 | 8 | 2
  RBC: Normal | 36 | 131 | 131 | 64
  RBC: Above | 0 | 1 | 0 | 2
  TP: Unknown | 0 | 0 | 0 | 0
  TP: Below | 0 | 0 | 0 | 0
  TP: Normal | 38 | 142 | 142 | 72
  TP: Above | 0 | 0 | 0 | 0
  WBC: Unknown | 0 | 3 | 3 | 3
  WBC: Below | 0 | 6 | 2 | 2
  WBC: Normal | 37 | 132 | 137 | 64
  WBC: Above | 1 | 1 | 0 | 3

ADVERSE EVENTS:
Time Frame: Solicited local/general symptoms: during the 7-day post-vaccination period (Days 0-6); Unsolicited AEs: during the 30-day post-vaccination period (Days 0-29); SAEs: during the entire study period (Day 0 - Month 14).
Arm/Group | Placebo Group | GSK1437173A Formulation 3 Group | GSK1437173A Formulation 2 Group | GSK1437173A Formulation 1 Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 2/73 | 0/149 | 1/150
Serious Adverse Events (participants affected / at risk) | 3/38 | 8/73 | 6/149 | 10/150
Other Adverse Events (participants affected / at risk) | 9/38 | 31/73 | 114/149 | 131/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=38) | GSK1437173A Formulation 3 Group (N=73) | GSK1437173A Formulation 2 Group (N=149) | GSK1437173A Formulation 1 Group (N=150)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus node dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pancreatic mass (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bile duct obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=38) | GSK1437173A Formulation 3 Group (N=73) | GSK1437173A Formulation 2 Group (N=149) | GSK1437173A Formulation 1 Group (N=150)
Chills (General disorders) | 0 (0) | 0 (0) | 3 (4) | 8 (10)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 27 (36) | 47 (66)
Fatigue (General disorders) | 7 (8) | 16 (20) | 52 (73) | 73 (101)
Gastrointestinal disorder (Gastrointestinal disorders) | 3 (3) | 5 (5) | 18 (22) | 17 (20)
Headache (Nervous system disorders) | 5 (6) | 11 (14) | 37 (50) | 57 (76)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 12 (16) | 49 (69) | 63 (93)
Pain (General disorders) | 3 (3) | 14 (17) | 104 (171) | 126 (220)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 18 (21) | 26 (33)
Swelling (General disorders) | 0 (0) | 3 (3) | 25 (29) | 24 (27)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.